CLINICAL TRIAL: NCT07198334
Title: The Effect of Daily Brief Whole-body Heat Exposures on Heat Acclimation and Its Decay
Brief Title: The Effect of Daily Brief Heat Exposures on Heat Acclimation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LithuanianSportsU-26
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat acclimation (Experimental)
  Interventions: Other: Heat acclimation

INTERVENTIONS:
Other: Heat acclimation — Passive heat acclimation was designed to induce adaptation in participants through 14 consecutive days of controlled 5-minute whole-body immersion in water at 45°C.

SUMMARY:
This study is the first to examine the effects of short passive heat exposure on heat acclimation (HA). Unlike traditional protocols requiring prolonged heat exposure, this study tests whether a daily 5-minute whole-body immersions at 45°C water repeated over two weeks can trigger adaptive responses, offering a potentially more accessible and time-efficient method for heat acclimation. This study aims to investigate whether brief, repeated passive heat exposure can induce HA in both female and male participants. It evaluates changes across physiological, biological, and psychological markers to determine the efficacy of this minimal-exposure protocol. It is hypothesized that such short, repeated immersions may be sufficient to elicit significant adaptive responses across key HA indicators.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-obese males and females aged 18 to 35 years with a body mass index between 18.5 and 29.9 kg/m².
* No participation in temperature manipulation programs (e.g., cold or heat acclimation) within the past three months.
* No engagement in excessive formal exercise.
* Female participants must have a regular menstrual cycle.

Exclusion Criteria:

* Current smokers.
* Fear of needles or blood.
* Use of medications or supplements that could affect study outcomes.
* History of neurological, cardiovascular, metabolic, or inflammatory diseases that could be aggravated by hot water exposure.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Dehydration (kg) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Dehydration (in kg) was assessed by calculating body mass loss (Tanita Body Composition Analyzer; USA) during heat exposure.
Heart rate (bpm) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Heart rate (in bpm) was recorded using a heart rate sensor with a chest strap (Polar, Finland).
Blood pressure (mmHg) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Systolic and diastolic blood pressure (in mmHg) was measured using with an automatic cuff monitor (Gentle+, Microlife, Switzerland).
Pulse pressure (mmHg) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Pulse pressure (in mmHg) was calculated by subtracting diastolic blood pressure from systolic blood pressure.
Rate of pressure production (AU) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Rate of pressure production (in AU) was calculated by multiplying heart rate , by systolic blood pressure.
Shivering/sweating (points) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  The shivering/sweating rate will be evaluated using 7-point scale. The rating of shivering/sweating range from 1 (heavily sweating) to 7 (vigorously shivering), with 4 being neutral.
Thermal comfort (points) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Thermal comfort will be evaluated using 4-point scale. The rating of thermal comfort range from 0 (neutral) to 3 (very uncomfortable).
Body temperature (°C) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Rectal temperature (in °C) was measured using a thermocouple (Rectal Probe, Ellab, Denmark) inserted to a depth of 12 cm past the anal sphincter, skin temperature (in °C) was measured with thermistors (Skin/Surface Probe, DM852, Ellab), and muscle temperature (in °C) was measured using a needle microprobe (MKA; Ellab).
Physiological strain index | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Physiological strain index (PSI) was used to indicate heat strain. PSI = 5 x (Tret - Tre0) x (39.5 - Tre0)^-1+ 5 x (HRt - HR0) x (180 - HR0)^-1, where rectal temperature (Tre) t and heart rate (HR) t are simultaneous measurements taken at the end of the heat exposure and Tre0 and HR0 are the initial measurements.
Oxygen consumption (mL/min/kg) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Oxygen consumption (in mL/min/kg) was measured using Cortex METALYZR® 3B, Leipcig, Germany).
Carbon dioxide output (mL/min/kg) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Carbon dioxide output (in mL/min/kg) was measured using Cortex METALYZR® 3B, Leipcig, Germany).
Carbon dioxide output (mL/min) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Carbon dioxide output (in mL/min) was measured using Cortex METALYZR® 3B, Leipcig, Germany).
Oxygen consumption (mL/min) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Oxygen consumption (in mL/min) was measured using Cortex METALYZR® 3B, Leipcig, Germany).
Respiratory quotient | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  The respiratory quotient was calculated by dividing the carbon dioxide output by the oxygen consumption. This ratio was used to assess substrate utilization. The values for fat is assumed as 0.7, for protein is assumed as 0.8 and for carbohydrate is assumed as 1.0.
Ventilation (L/min) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Ventilation (in L/min) was measured using Cortex METALYZR® 3B, Germany).
Tidal volume (L) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Tidal volume (in L) was measured using Cortex METALYZR® 3B, Germany).
Breathing frequency (t/min) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Breathing frequency (t/min) was measured using Cortex METALYZR® 3B, Germany).

SECONDARY OUTCOMES:
Height (cm) | During enrollment
  Height (in cm) was measured using a Harpenden anthropometer set (Holtain Ltd, UK).
Body mass and body composition (kg) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Body mass and composition (in kg) was evaluated using Tanita Body Composition Analyzer (USA).
Body mass index (kg/m^2) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Body mass index (in kg/m^2) will be defined as the body mass divided by the square of the body height.
Body composition (%) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Body composition (in %) was evaluated using Tanita Body Composition Analyzer (USA).
Maximal oxygen consumption (in mL/min/kg) | During enrollment
  Maximal oxygen consumption (VO2max) (in mL/min/kg) was defined through a maximal incremental exercise test conducted on an electromechanically braked cycling ergometer (Ergometrics-800S; Ergoline Medical Measurement Systems, Germany) and was measured on a breath-by-breath basis using a stationary MetaLyzer® 3B spiroergometry system (Cortex Biophysik GmbH, Germany).
Prolactin (ng/mL) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Serum prolactin (in ng/mL) was measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria).
17beta-estradiol (pg/mL) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Serum 17beta-estradiol (in pg/mL) was measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria).
Progesterone (ng/mL) | From enrollment to the end of deacclimation (one month after the 14-day heat acclimation period).
  Serum progesterone (in ng/mL) was measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria).

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided